CLINICAL TRIAL: NCT03469830
Title: The Effectiveness of a Smart Scar Care Pad and Pressure Therapy Versus Pressure Therapy in Hypertrophic Scar Management: a Pilot Study
Brief Title: The Development and Application of "Scar-care" Padding on Management of Hypertrophic Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140618002-01
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cicatrix, Hypertrophic; Rehabilitation
Keywords: insert; pressure therapy; silicone gel
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Polymorphism, Single-Stranded Conformational

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subjects and the analyser of the data were blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSCP & SPMS (Experimental): The smart scar care pad (SCCP):
  The SCCP is a newly invented insert material that can maximise treatment outcomes via enhanced compression and occlusion. The wearing regime for SCCP is 4 hours a day for the first day, with 2-hour increments added every other day until the total wearing time reached 23 hours. SSCP was cleaned twice a day for hygienic reasons.
  The smart pressure monitored suit(SPMS):
  The SPMS is a type of custom-made pressure garment. SPMS was used 23 hours a day and only removed when showering.
  Interventions: Other: SSCP; Other: SPMS
- SPMS (Active Comparator): The smart pressure monitored suit(SPMS):
  The SPMS is a type of custom-made pressure garment. SPMS was used 23 hours a day and only removed when showering.
  Interventions: Other: SPMS

INTERVENTIONS:
Other: SSCP — Insert
  Other Names: The Smart Scar Care PAd
  Arms: SSCP & SPMS
Other: SPMS — Pressure therapy
  Other Names: The Smart Pressure Monitored Suit

SUMMARY:
This study explores the smart scar care pad's potential therapeutic effect in treatment hypertrophic scar while elucidating the adverse effects if there is any. Half of the participant receives traditional treatment of pressure garment and the other half receives the smart scar care pad together with pressure garment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Hypertrophic Scar(HS);
2. the HS had a total Vancouver Scar Scale (VSS) score of 4 or higher and the score of each item equal to or greater than 1;
3. subjects age between 20 and 70 years, cooperative, and good compliance with treatment.

Exclusion Criteria:

1. the HS area had an open wound or infection;
2. the HS had been treated with steroid injections or other intervention (such as traditional Chinese medicine or laser therapy) before the study; or
3. the patient had a medical condition that might affect wound healing (e.g., diabetes mellitus or another serious medical problem).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Change of Scar Pliability measured by the DermaLab Combo | baseline and 6 weeks
  Scar pliability is represented by the Young's modulus measured by the elasticity measurement of the DermaLab Combo

SECONDARY OUTCOMES:
Change of Scar Thickness measured by the diagnostic ultrasound system | baseline and 6 weeks
  Scar thickness is measured by the diagnostic ultrasound system
Change of Scar Pigmentation measured by the DermaLab Combo | baseline and 6 weeks
  Scar pigmentation is represented by the melanin score generated by the color probe of the DermaLab Combo. The range of the score is 0-100, where a higher score indicates a higher melanin content.
Change of Scar Vascularity measured by the DermaLab Combo | baseline and 6 weeks
  Scar vascularity is represented by the erythema score measured by the color probe of the DermaLab Combo. The range of the score is 0-100, where a higher score indicates a more erythematic situation.
Occurrence of blistering | up to 6 weeks
  Occurence of blistering is observed and reported by research staff
Occurrence of skin breakdown | up to 6 weeks
  Occurence of skin breakdown is observed and reported by research staff
Occurrence of rash | up to 6 weeks
  Occurence of rash is observed and reported by research staff